CLINICAL TRIAL: NCT05202197
Title: Smart Cupboard-based System for Memory Assessment in Alzheimer's Patients
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Guillermo Palacios, Principal Investigator, Universidad de Zaragoza
Other Study IDs: PI21/326
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer Disease; Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Alzheimer´s patients
  Interventions: Other: Smart cupboard

INTERVENTIONS:
Other: Smart cupboard — Development of a memory task with the help of a smart cupboard

SUMMARY:
The main objective of the research is to create a tool that can make a good diagnosis of cognitive abilities in Alzheimer's patients. As a secondary objective, the investigators intend to examine both the percentage of correct answers and the response times and see their relationship with age, gender, sex, months since the onset of the disease and years of training.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years.
2. Provide signed informed consent.
3. Have the ability to understand the study.

Exclusion Criteria:

Having any physical or medical problem that prevents or advises them not to stand upright, in a bipedal position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community dwelling Alzheimer's patients who attend the Alzheimer's and dementia center in Teruel on a regular basis.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Accuracy response. | 60 minutes
  Number of successes / failures on the total of questions
Reaction time | 60 minutes
  Defined as the time it takes the subject to answer each of the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Teruel, Spain

IPD SHARING:
Plan to Share IPD: No